CLINICAL TRIAL: NCT00663481
Title: A Single Dose, Within Subject, 3 Period, Pharmacokinetic Bridging Study of CoFactor Formulations and of Leucovorin Administered Intravenously in Healthy, Adult Subjects.
Brief Title: A Clinical Trial of CoFactor Formulations and Leucovorin Administered Intravenously in Healthy, Adult Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Jeff Stewart, MBA, ADVENTRX Pharmaceuticals, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CoFactor 510-20
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Adults
Keywords: CoFactor; ANX-510
MeSH Terms: interventions — 5,11-methenyltetrahydrohomofolate; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): CoFactor
  Interventions: Drug: CoFactor
- 2 (Experimental): CoFactor
  Interventions: Drug: CoFactor
- 3 (Active Comparator): Leucovorin
  Interventions: Drug: Leucovorin

INTERVENTIONS:
Drug: CoFactor
  Other Names: ANX-510
  Arms: 1; 2
Drug: Leucovorin
  Arms: 3

SUMMARY:
The purpose of this study is to determine the safety and tolerability of CoFactor in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 18-65 inclusive at screening.
* Subject has to agree to practice abstinence or medically accepted contraception and not to participate in sperm donation or in vitro fertilization.
* Body Mass Index in the range of 18 to 30 kg/m2 and body weight of 45 to 95 kg.
* Subject must be healthy as determined by the investigator on the basis of screening evaluations.
* Subject must be nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the in-clinic stay.

Exclusion Criteria:

* Presence of clinically significant illness within 21 days prior to dosing, viral or bacterial infection, or documented drug allergies that may affect subject's safety during the study.
* Laboratory or clinical evidence suggestive of disease.
* Clinically significant or predisposing disorder that may interfere with the absorption, distribution, metabolism and/or excretion of drugs.
* History of drug abuse within 1 year of dosing and/or admitted alcohol abuse or history of alcohol use that may interfere with the ability to comply.
* Pregnant, lactating, or positive pregnancy test.
* Clinically significant electrocardiogram abnormalities.
* History of positive test for hepatitis B or C, or HIV.
* Positive findings of urine narcotic screen.
* History of drug allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of CoFactor formulations in healthy adult subjects.

SECONDARY OUTCOMES:
To measure the 5,10 methylenetetrahydrofolic acid levels after CoFactor and leucovorin administration

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — Parexel International - Baltimore CPRU
Locations (1):
- Parexel International - Baltimore CPRU, Baltimore, Maryland, United States